CLINICAL TRIAL: NCT06176274
Title: The Effect of Pre-Operative Prehabilitation Program on Postoperative Recovery in Women With Gynecological Cancer
Brief Title: Pre-Operative Prehabilitation Program Women With Gynecological Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Hilal Evgin, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IstanbulUC-LEE-HE-01
Record Dates: First submitted 2023-12-10; First posted 2023-12-19 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-06

CONDITIONS: Gynecologic Cancer; Prehabilitation
Keywords: Prehabilitation; cancer; Gynecologic cancer; nursing
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: a randomized trial with experimental design with pre-test post-test control group
Who Masked: Participant, Care Provider
Masking Description: the experimental group will receive care through the prehabilitation program, while the control group will receive standard nursing care. participants will not know which group they are in.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the experimental group (Experimental): a prehabilitation program will be applied before the surgery.
  Interventions: Other: Prehabilition program
- The Control Group (No Intervention): he will receive standard nursing care procedure.

INTERVENTIONS:
Other: Prehabilition program — this program includes nutrition, physical activity, medical optimization and psychological support interventions.As a practice, the prehabilitation program (according to the surgery program) is planned in the preoperative period between 2-4 weeks Dec. it will be applied for 4 weeks before surgery. the first meeting is scheduled for 40 minutes. the program compliance process will be monitored by phone weekly. postoperative recovery and functional capacity measurements will be performed.
  Arms: the experimental group

SUMMARY:
The aim of this study is to determine the effect of the prehabilitation program applied to postmenopausal women diagnosed with gynecological cancer before surgery on postoperative recovery, planned as a randomized study with an experimental design with a pre-test post-test control group.

DETAILED DESCRIPTION:
The aim of prehabilitation programs is to eliminate intraoperative complications by increasing the functional capacity and metabolic reserves of patients before surgical treatment and to accelerate recovery in the postoperative period. In addition, it helps the patient to maximize the existing capacity of the patient before the surgery, to know what will happen at each stage of the treatment to be applied to the patient, to feel better physically and spiritually and to understand the roles and responsibilities of the individual care of the patient, as well as making a significant contribution to the positive results of the operation. It is to provide exercise, psychological support, nutritional counseling and optimization of the underlying conditions by stopping negative health behaviors. There are non-eliminable criteria such as age, gender, comorbid diseases before surgery, as well as modifiable factors such as the regulation of the patients nutrition, ensuring psychological well-being, quitting smoking. In particular, some factors directly affect the state of well-being during the perioperative period. Thus, surgeries become safer.As a practice, the prehabilitation program (according to the surgery program) is planned in the preoperative period between 2-4 weeks Dec. Participants who do not comply with the program will be excluded from the sample

ELIGIBILITY:
Inclusion Criteria:

* Patients who are not stage 4 in preoperative evaluation
* Who volunteered to participate in the study
* 6 months have passed since the last treatment (Chemoretapy, Radiotherapy)
* Women who do not have Turkish literacy problems
* Women aged 50 and older who are in the postmenopausal period
* Patients who are scheduled for abdominal surgery

Exclusion Criteria:

* High-risk comorbid diseases such as COPD, heart failure
* Physical and mental conditions that will interfere with nutrition and exercise
* Those with orthopedic and neuromuscular diseases
* Those who are scheduled for surgery by laparoscopic/laparotomic method
* Those who cannot adapt to the program during the preoperative period
* Women who are too depressed during preoperative evaluation

Min Age: 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
the Quality of Recovery QoR-15 | 6 weeks
  The scale is based on the assumption that the higher the score, the better the quality of improvement when measuring between 0 and 150 points. The scale is based on the assumption that the higher the score, the better the quality of Deceleration.
functional capacity 6MWT | 10 weeks
  6MWT has also been used to determine the functional status of patients . During the test, a standardized protocol is followed by walking on a flat floor for 6 minutes. It is a self-paced test and is a repeatable, cheap and easy test (unlike the increasingly brisk walking tests that require intervention).
day of hospital stay | 1 weeks
  the length of hospital stay
the WHODASS proficiency scale | 1 weeks
  the WHODASS proficiency scale will be used. It is useful for a brief assessment of the overall functionality.

CONTACTS AND LOCATIONS:
Overall Officials: hilal Evgin, Phd Student, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Prof Dr Cemil Taşçıoğlu City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No